CLINICAL TRIAL: NCT05357014
Title: Evaluation Of Cardiac Function In Children 0n Regular Heamodialysis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Fatma Ahmed Sahy, resident doctor at pediateric department sohag university hospital, Sohag University
Other Study IDs: Soh-Med-22-04-10
Record Dates: First submitted 2022-04-17; First posted 2022-05-02 (Actual); Last update posted 2022-05-02 (Actual); Status verified 2022-04

CONDITIONS: Children on Regular Heamodialysis
MeSH Terms: interventions — Echocardiography

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: echocardiography — evaluation of cardiac function hn children on regular heamodialysis by echocardiography

SUMMARY:
Cardiovascular disease (CVD) is considered as the predominant cause of mortality and morbidity in chronic kidney disease (CKD) patients .

* Left ventricular diastolic and systolic dysfunction and left ventricular hy pertrophy (LVH) contribute to the increased cardiovascular mortality rate in these patients .Such changes have been observed in young adults and children on prolonged dialysis
* The cardiovascular mortality and morbidity are seen in earlier stages of CKD, and the risk is increased by multiple risk factors such as sodium and fluid retention,hypertension, anemia, inflammation and hyperparathyroidism .
* Left ventricular hypertrophy is a common finding in CKD patients [8] and its severity increases with increasing severity of CKD . Initially, LVH is discussed as a physiological response to volume and pressure overload. However, sustained overload in combination with CKD associated risk factors may result in maladaptive LVH characterized by structural changes in the myocardium (calcification, fibrosis and collagen accumulation), resulting in diastolic and systolic dysfunction .
* Causes of LV diastolic dysfunction are impaired active LV relaxation or decreased LV compliance.These changes are reflected in low diastolic volume for a given diastolic pressure, meaning reduced passive LV filling .
* Changes in cardiac structure and function are common among the patients with chronic kidney disease undergoing hemodialysis. As early as 1827, Richard Bright drew attention to the common presence of left ventricular hypertrophy and thickening of the aortic wall in the patients with end-stage renal disease (ESRD).
* Cardiovascular (CV) disease is the leading cause of mortality in the childhood renal replacement therapy population with long-term observational studies reporting 40-45% deaths attributable to CV disease , increasing to 57% when stratified to haemodialysis patients only . In children with CKD, left ventricular hypertrophy (LVH) is common and occurs early in the disease process with reported prevalence up to 65% and increasing to 82% in those on haemodialysis .

  * The present study stresses the importance of echocardiography as the gold standard for the diagnosis of cardiac disease in pediatric patients under maintenance HD as a high-risk population for cardiac diseases.

ELIGIBILITY:
Inclusion Criteria:

* All patients (2-18) years were undergoing regular HD, who were started on dialysis when GFR was ≤15 mL/min/1.73 m 3 three times per week, with each dialysis session lasting for 3-4 h.

Exclusion Criteria:

* Patients of primary cardiac diseases (e.g., congenital or rheumatic heart disease, cardio- myopathy).

Ages: 2 Years to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: All patients (2-18) years were undergoing regular HD, who were started on dialysis when GFR was ≤15 mL/min/1.73 m 3 three times per week, with each dialysis session lasting for 3-4 h.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2022-05 (Estimated); Primary Completion 2023-05 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
Left ventricular mass (LVM). | one year
  Left ventricular mass (LVM) will be calculated using the measurements obtained by two-dimensional directed M-mode echocardiography according to the American Society of Echocardiography (ASE) criteria . Indexed LVM (LVMI) will be calculated by dividing the LVM by height raised to a power of 2.7 (g/m2.7) using the formula devised by De Simone et al(De Simone G1992)
Diastolic function . | one year
  Diastolic function will be assessed by both Doppler echocardiography and tissue Doppler imaging. Early mitral inflow velocity (E), and late mitral inflow velocity (A) will be measured by Doppler echocardiography. Early (e) and late (a') peak mitral annular velocities will be measured at the medial and lateral mitral annulus using tissue Doppler. The e'/a' ratio at both annuli will be calculated. The peak early mitral annular velocity (E') will be computed as the average of the velocities at the medial and lateral annuli. Using these measurements, the ratio of Doppler-derived peak early mitral inflow velocity to tissue Doppler-derived peak early mitral annular velocity (E/E'ratio) will be calculated.
The left ventricular myocardial performance index (MPI). | one year
  The left ventricular myocardial performance index (MPI), a global index of systolic and diastolic function, will be defined as the sum of isovolumic relaxation time and isovolumic contraction time divided by ejection time.

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Al-Biltagi M, Tolba OA, ElHafez MA, Abo-Elezz AA, El Kady EK, Hazza SM. Oxidative stress and cardiac dysfunction in children with chronic renal failure on regular hemodialysis. Pediatr Nephrol. 2016 Aug;31(8):1329-39. doi: 10.1007/s00467-016-3314-8. Epub 2016 Mar 18. PMID 26993814
- [Background] Yeh HM, Lin TT, Yeh CF, Huang HS, Chang SN, Lin JW, Tsai CT, Lai LP, Huang YY, Chu CL. Biomarkers and echocardiography for evaluating the improvement of the ventricular diastolic function after surgical relief of hydronephrosis. PLoS One. 2017 Nov 21;12(11):e0188597. doi: 10.1371/journal.pone.0188597. eCollection 2017. PMID 29161313
- [Background] Collins AJ, Foley RN, Chavers B, Gilbertson D, Herzog C, Johansen K, Kasiske B, Kutner N, Liu J, St Peter W, Guo H, Gustafson S, Heubner B, Lamb K, Li S, Li S, Peng Y, Qiu Y, Roberts T, Skeans M, Snyder J, Solid C, Thompson B, Wang C, Weinhandl E, Zaun D, Arko C, Chen SC, Daniels F, Ebben J, Frazier E, Hanzlik C, Johnson R, Sheets D, Wang X, Forrest B, Constantini E, Everson S, Eggers P, Agodoa L. 'United States Renal Data System 2011 Annual Data Report: Atlas of chronic kidney disease & end-stage renal disease in the United States. Am J Kidney Dis. 2012 Jan;59(1 Suppl 1):A7, e1-420. doi: 10.1053/j.ajkd.2011.11.015. No abstract available. PMID 22177944
- [Background] Mitsnefes MM. Cardiovascular disease in children with chronic kidney disease. J Am Soc Nephrol. 2012 Apr;23(4):578-85. doi: 10.1681/ASN.2011111115. Epub 2012 Mar 1. PMID 22383696